CLINICAL TRIAL: NCT06859658
Title: Développement et Validation d'un Biomarqueur en IRM Fonctionnelle de la Dysfonction Des Petits Vaisseaux cérébraux Dans la Maladie de CADASIL
Brief Title: Development and Validation of a Functional MRI Biomarker of Cerebral Small Vessel Dysfunction in CADASIL
Acronym: fMRI BioSVD
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240772
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: CADASIL
Keywords: fMRI; Cerebral Small Vessel Diseases; Neurovascular coupling; CADASIL; Biomarkers
MeSH Terms: conditions — CADASIL; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group
  Interventions: Radiation: Functional MRI at 3T
- CADASIL patients with no disability or significant cognitive deficit
  Interventions: Radiation: Functional MRI at 3T
- CADASIL Patients with mild to moderate disability or with a moderate cognitive deficit
  Interventions: Radiation: Functional MRI at 3T

INTERVENTIONS:
Radiation: Functional MRI at 3T — At inclusion
  Groups: Control group
Radiation: Functional MRI at 3T — At inclusion and at 2 years for CADASIL patients without severe disability (mRS<4)
  Groups: CADASIL patients with no disability or significant cognitive deficit
Radiation: Functional MRI at 3T — At inclusion and at 2 years for CADASIL patients without severe disability (mRS<4)
  Groups: CADASIL Patients with mild to moderate disability or with a moderate cognitive deficit

SUMMARY:
Cerebral small vessel diseases (cSVD) are diseases of brain tissue involving vessels (arterioles or capillaries) with a diameter of less than 400 microns. Within this group, CADASIL (Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy) is the most common familial form. CADASIL is due to mutations in the NOTCH3 gene located on chromosome 19. It is considered a unique model for the study of cSVD. CADASIL begins between the ages of 20 and 40, with the appearance of cerebral white matter hyper-signals visible on MRI. Before the age of 30, patients are usually asymptomatic. To date, there are no available treatments. To test new therapeutic approaches, we need biomarkers that are robust and sensitive enough to assess the effects of these treatments at an early stage of cSVD and over a relatively short period of time.

An ideal monitoring biomarker should be repeatedly and safely usable, easily accessible, accurate, reproducible and sensitive to disease progression or pharmacological intervention.

Alterations in neurovascular coupling (NVC) have been recognized as one of the earliest functional alterations occurring during cSVD. Cerebral functional magnetic resonance imaging (fMRI) is a brain imaging technique that measures the activity of brain areas in vivo by detecting local changes in blood flow. An important advantage of blood oxygen level-dependent functional MRI is that it enables the NVC to be probed in vivo, safely and repeatedly in humans.

Our central hypothesis is that functional MRI can provide such a biomarker for monitoring CNV disease progression in vivo using a dedicated fMRI protocol that can be used on a clinical MRI scanner, is reproducible and varies according to the severity of brain MRI lesions and/or clinical manifestations in CADASIL. A functional imaging study coupled with electroencephalogram has already revealed changes in the hemodynamic response to visual or motor stimuli in patients at the early stage of the disease. This study is exploring new imaging protocols to focus on the purest vascular response.

ELIGIBILITY:
Inclusion criteria :

For CADASIL patients

* Age between 18 and 80 at the time of inclusion
* Diagnosis confirmed by detection of a pathogenic mutation in the NOTCH3 gene characteristic of CADASIL.
* Beneficiaries of a health insurance.
* Written consent.

For controls:

* Age between 18 and 80 at the time of inclusion
* Beneficiary of a health insurance.
* Written consent

Exclusion criteria :

For patients

* Contraindication to MRI examination
* Disability: Rankin score ≥ 4
* Moderate to severe dementia according to DSM 5 criteria or MMSE score ≤ 19
* Person covered by articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the French Public Health Code, defined by :

  * Pregnant, parturient or breast-feeding woman
  * Person deprived of liberty by judicial or administrative decision.
  * Persons hospitalized without consent and not under legal protection, and persons admitted to a health or social establishment for purposes other than research.
  * Minor
  * Person of full age subject to a legal protection measure (guardianship, curatorship or safeguard of justice), person of full age unable to give consent and not subject to a protection measure.
* Person subject to a period of exclusion for another research project

For controls :

* Contraindication to MRI examination
* Known cognitive complaint or deficit
* Presence of significant disability (mRS >1)
* Focal neurological motor, sensory or visual deficit on clinical examination that may impair visual or motor stimulation tests
* History of neurological or psychiatric disease
* History of migraine attacks with aura
* Vascular history (known disease of peripheral arteries, heart or brain)
* Known or treated diabetes
* Known or treated hypercholesterolemia
* Known or treated hypertension
* Active smoking or smoking cessation within the last year
* Regular alcohol consumption corresponding to > 2 glasses/day for men and 1 glass/day for women in wine equivalent
* Treatment likely to interfere with neurovascular coupling (in particular any treatment with non-steroidal anti-inflammatory drugs, psychotropic drug(s), antihypertensive drug(s) or statins)
* Person covered by articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the French Public Health Code, defined by :

  * Pregnant, parturient or breast-feeding woman
  * Person deprived of liberty by judicial or administrative decision
  * Persons hospitalized without consent and not under legal protection, and persons admitted to a health or social institution for purposes other than research.
  * Minor
  * Person of full age subject to a legal protection measure (guardianship, curatorship or safeguard of justice), person of full age unable to give consent and not subject to a protection measure.
  * Person subject to a period of exclusion for another research project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a known mutation in the NOTCH3 gene
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Variation in BOLD response | At inclusion
  Variation in BOLD response on functional MRI during short-duration visual stimuli (area under the curve) and parameters derived from this response curve at the calcarine scissure For all patients and controls
Variation in BOLD response | At 2 years
  Variation in BOLD response on functional MRI during short-duration visual stimuli (area under the curve) and parameters derived from this response curve at the calcarine scissure For CADASIL patients

SECONDARY OUTCOMES:
Correlations between parameters derived from the response curve and age | Up to 2 years
Correlations between parameters derived from the response curve and gender | Up to 2 years
Correlations between parameters derived from the response curve and cardiovascular risk factors | Up to 2 years
Correlations between parameters derived from the response curve and modified Rankin score | Up to 2 years
Correlations between parameters derived from the response curve and stroke frequency | Up to 2 years
Correlations between parameters derived from the response curve and stroke number | Up to 2 years
Correlations between parameters derived from the response curve and total brain volume | Up to 2 years
Correlations between parameters derived from the response curve and cerebral parenchymal fraction | Up to 2 years
Correlations between parameters derived from the response curve and normalized WMH (White matter hyperintensity)volume | Up to 2 years
Correlations between parameters derived from the response curve and number of microbleeds | Up to 2 years
Correlations between parameters derived from the response curve and number of lacunae | Up to 2 years

IPD SHARING:
Plan to Share IPD: Undecided